CLINICAL TRIAL: NCT02361749
Title: Comparative Study Between Botulinum Toxin Injection and Myectomy in Treatment of Idiopathic Constipation in Children
Brief Title: Botulinum Toxin Injection Versus Anal Myectomy in Management of Idiopathic Constipation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Elfiky, MD, Lecturer of Pediatric Surgery, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIUNIPEDSURG-CR2; PACTR201408000857349 (Other: PACTR)
Record Dates: First submitted 2015-01-09; First posted 2015-02-12 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Chronic Idiopathic Constipation; Functional Constipation
MeSH Terms: interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myectomy group (Active Comparator): Subjects will undergo anal myectomy for their anal sphincter.
  Interventions: Procedure: Anal Myectomy
- Botox Group (Active Comparator): Subjects will undergo Botulinum toxin injection into their anal sphincter.
  Interventions: Drug: Botulinum Toxin

INTERVENTIONS:
Drug: Botulinum Toxin — Injection of Botulinum toxin under general anesthesia. Four injections will be given into the anal sphincter into the four quadrants in one session.
  Other Names: Botox
  Arms: Botox Group
Procedure: Anal Myectomy — Longitudinal anal myectomy will be performed under general anesthesia as a day case.
  Arms: Myectomy group

SUMMARY:
Chronic idiopathic constipation is most common cause of Constipation in childhood with numerous cases in Egypt. Numerous conservative measures were tried but many fail. Surgical options include Longitudinal Myectomy of the muscle or injection of Botulinum toxin. Objectives: Comparative study between Botulinum toxin injection and Myectomy in treatment of Idiopathic Constipation

DETAILED DESCRIPTION:
Functional constipation (chronic idiopathic constipation) is most common cause of constipation in pediatric age group. Many cases try conservative treatment but fail to respond. These cases are treated by surgical longitudinal myectomy of the anal sphincter. Now, there have been many trials of trying injection of botulinum toxin to relax the sphincter as a treatment of functional/idiopathic constipation.

In this study, the investigators will compare the results of botulinum toxin injection versus surgical myectomy to treat functional/idiopathic constipation in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with Idiopathic constipation

Exclusion Criteria:

* Hirschsprung's disease or Anorectal malformations

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Absence of insufficient Rome III Diagnostic criteria (0-1 criterion) | 2 years
  Rome III Diagnostic criteria for chronic idiopathic constipation include two or more of the following in a child with a developmental age of at least 4 years:
  1. Two or fewer defecations in the toilet per week
  2. At least one episode of fecal incontinence per week
  3. History of retentive posturing or excessive volitional stool retention
  4. History of painful or hard bowel movements
  5. Presence of a large fecal mass in the rectum
  6. History of large diameter stools which may obstruct the toilet
  Outcome measure for Curing Chronic idiopathic constipation is denoted by absence of insufficient criteria (0-1 criterion) to diagnose Chronic idiopathic constipation after receiving corresponding arm of the study.

SECONDARY OUTCOMES:
Decrease in Rome III Diagnostic criteria score | 2 years
  Rome III Diagnostic criteria for chronic idiopathic constipation include two or more of the following in a child with a developmental age of at least 4 years:
  1. Two or fewer defecations in the toilet per week
  2. At least one episode of fecal incontinence per week
  3. History of retentive posturing or excessive volitional stool retention
  4. History of painful or hard bowel movements
  5. Presence of a large fecal mass in the rectum
  6. History of large diameter stools which may obstruct the toilet
  Outcome measure for improving Chronic idiopathic constipation is denoted by giving each case a 6-point score system based on Chronic idiopathic constipation diagnostic criteria. Improvement is denoted by decrease in diagnostic criteria score after receiving corresponding arm of the study. The decrease is assessed, analyzed and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Seoudi, Principal Investigator — Cairo University
Locations (1):
- Cairo University Pediatric Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
WOFAPS 2016

REFERENCES:
- [Background] Keshtgar AS, Ward HC, Sanei A, Clayden GS. Botulinum toxin, a new treatment modality for chronic idiopathic constipation in children: long-term follow-up of a double-blind randomized trial. J Pediatr Surg. 2007 Apr;42(4):672-80. doi: 10.1016/j.jpedsurg.2006.12.045. PMID 17448764
- [Background] Irani K, Rodriguez L, Doody DP, Goldstein AM. Botulinum toxin for the treatment of chronic constipation in children with internal anal sphincter dysfunction. Pediatr Surg Int. 2008 Jul;24(7):779-83. doi: 10.1007/s00383-008-2171-3. Epub 2008 Apr 29. PMID 18443801
- [Background] Hata Y, Sasaki F, Uchino J. Sphincteromyectomy and sphincteroplasty in chronic constipation with megarectum. J Pediatr Surg. 1988 Feb;23(2):141-2. doi: 10.1016/s0022-3468(88)80143-x. PMID 3343649
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553